CLINICAL TRIAL: NCT05423483
Title: Developing an Intervention to Promote Lethal Means Safety in Suicidal Adolescents: Randomization
Brief Title: Developing an Intervention to Promote Lethal Means Safety in Suicidal Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Beth Kennard, Professor of Psychiatry, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU-2022-0396
Record Dates: First submitted 2022-05-31; First posted 2022-06-21 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Text Message Intervention (Experimental): Parents in the intervention arm will receive text message reminders to restrict lethal means for 6 months.
  Interventions: Behavioral: Safe Home Text Message Reminders
- Treatment as Usual (No Intervention): Parents in the treatment as usual group will not receive the text message intervention.

INTERVENTIONS:
Behavioral: Safe Home Text Message Reminders — Text messages sent 2x a week with reminders to keep lethal means restricted and surveys of lethal means practices that serve as a prompt to adhere to suggested restriction measures.
  Arms: Text Message Intervention

SUMMARY:
Study Objective: to develop a phone-based intervention to aid parents of suicidal adolescents to adhere to lethal means safety.

Lethal means counseling is the practice of educating patients and their families about limiting access to items that can be used to attempt suicide. Though lethal means counseling is standard practice in treating suicidal patients, there is little experimental literature related to its utilization across different providers and its efficacy. Further, there is a significant gap in the literature on lethal means counseling as it relates to adolescents. The proposed project will investigate a novel text message-based intervention aimed to promote lethal means safety.

DETAILED DESCRIPTION:
Participants will be adolescents (age 12-17) who are currently enrolled in the SPARC IOP for a recent suicide attempt or significant suicidal ideation with a plan or intent and their parents or legal guardians. SPARC clinical staff will identify patients and parents who would be eligible based on inclusion/exclusion criteria provided to them. If the family is interested, the study staff will be on hand to present the study and collect informed assent from patients and consent from parent(s).

Investigators will enroll up to 120 pairs of parents and teens receiving care at the SPARC clinic. Investigators will utilize a Children's Health HIPAA compliant texting services to send prompts to the parents of the teens. Phase I of the study was approved in STU-2020-0100 in which the team developed interviews and data collection guides. In Phase II, approved in STU-2021-0658, the team is conducting pilot testing of the intervention to determine if parents find it useful. In this study, Phase III, investigators will randomize the families into two groups: the first being the treatment as usual (TAU) group (N = 60) and the second being the intervention group (N = 60). Parents and guardians in the control group will not receive the text-based intervention. In the intervention group, parents of teens currently enrolled in the SPARC program will enroll in and receive text-based reminders (safety prompts and questionnaire) to adhere to lethal means safety practices twice a week, serving as an intervention to increase adherence to lethal means safety. Data will be collected at 4 time points: SPARC intake, SPARC discharge, 1 month following SPARC discharge, and 6 month following SPARC discharge. At 1-month and 6-month follow up, parents will complete Client Satisfaction Questionnaire regarding satisfaction with the intervention, a brief measure of family functioning, and a brief measure of parental-self efficacy in the context of their child's suicidality. Additionally, at 1-month and 6-month follow up, adolescents will complete questionnaires regarding their access to lethal means in the time frame and measures of suicidality and symptomatology. All 1-month and 6-month questionnaires will be completed by families digitally or over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Proficiency in spoken and written English
* Own cell phone that has internet capabilities
* Adolescent participants are patient's at Children's Health SPARC IOP (ages 12-17)
* Adult participants are parents and/or legal guardians of adolescent participants (ages 18+)

Exclusion Criteria:

* Non-English speaking

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Adolescent suicidal behavior | 6 months
  Adolescent suicidal behavior will be measured by Columbia Suicide Severity Rating Scale (C-SSRS) which is used to measure suicidal thoughts and behaviors in Investigational New Drug (IND) studies. The C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent).
Parent satisfaction as measured by CSQ-8 | 6 months
  Parent satisfaction will be measured by Client Satisfaction Questionnaire (CSQ-8) which is a self report measure of satisfaction with health and behavioral services received. The CSQ-8 is measured on a four point Likert scale from 1 "Quite Dissatisfied" to 4 "Very Satisfied." Scores range from 8-32, with higher values indicating higher satisfaction
Parent suicide prevention self efficacy as measured by parent suicide prevention self efficacy scale | 6 months
  Parent suicide prevention self efficacy is measured by parent suicide prevention self efficacy scale which measures parent's confidence on a scale of 0 (not at all confident) to 10 (completely confident)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Health, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No